CLINICAL TRIAL: NCT00532298
Title: Non-Inferiority of GlaxoSmithKline Biologicals' Influenza Vaccine (GSK576389A) 1 Container Over 2 Container Presentation in Adults Aged 65 Years and Over
Brief Title: Non-Inferiority of Various GSK Bio's Influenza Vaccine Presentations in Adults Aged 65 Years and Over
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 110620
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Results first posted 2012-05-22 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2016-11

CONDITIONS: Influenza
Keywords: Fluarix; Influenza Infection; GSK Biologicals' influenza vaccine GSK576389A
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (6):
- GSK576389A- 2006/2007 Season - 1 container Group (Experimental): Subjects aged ≥ 65 years received adjuvanted influenza vaccine GSK576389A for the Northern Hemisphere 2006/2007 influenza season presented in 1 container.
  Interventions: Biological: GSK Bio's influenza vaccine GSK576389A [NH 2006/07 season]
- GSK576389A - 2006/2007 Season - 2 containers Group (Experimental): Subjects aged ≥ 65 years received adjuvanted influenza vaccine GSK576389A for the Northern Hemisphere 2006/2007 influenza season presented in 2 containers.
  Interventions: Biological: GSK Bio's influenza vaccine GSK576389A [NH 2006/07 season]
- Fluarix 2006/2007 Season Group (Active Comparator): Subjects aged ≥ 65 years received a single dose of Fluarix vaccine formulation recommended for the Northern Hemisphere 2006-2007 influenza season.
  Interventions: Biological: Fluarix [NH 2006/07 season]
- GSK576389A - 2007/2008 Season - 1 container Group (Experimental): Subjects aged ≥ 65 years received adjuvanted influenza vaccine GSK576389A for the Northern Hemisphere 2007/2008 influenza season presented in 1 container.
  Interventions: Biological: GSK Bio's influenza vaccine GSK576389A [NH 2007/08 season]
- GSK576389A - 2007/2008 Season - 2 containers Group (Experimental): Subjects aged ≥ 65 years received adjuvanted influenza vaccine GSK576389A for the Northern Hemisphere 2007/2008 influenza season presented in 2 containers.
  Interventions: Biological: GSK Bio's influenza vaccine GSK576389A [NH 2007/08 season]
- Fluarix 2007/2008 Season Group (Active Comparator): Subjects aged ≥ 65 years received a single dose of Fluarix vaccine formulation recommended for the Northern Hemisphere 2007-2008 influenza season.
  Interventions: Biological: Fluarix [NH 2007/08 season]

INTERVENTIONS:
Biological: GSK Bio's influenza vaccine GSK576389A [NH 2006/07 season] — Single dose, intramuscular injection, GSK Bio's influenza vaccine GSK576389A formulation recommended for the Northern Hemisphere 2006-2007 influenza season.
  Arms: GSK576389A - 2006/2007 Season - 2 containers Group; GSK576389A- 2006/2007 Season - 1 container Group
Biological: GSK Bio's influenza vaccine GSK576389A [NH 2007/08 season] — Single dose, intramuscular injection, GSK Bio's influenza vaccine GSK576389A formulation recommended for the Northern Hemisphere 2007-2008 influenza season.
  Arms: GSK576389A - 2007/2008 Season - 1 container Group; GSK576389A - 2007/2008 Season - 2 containers Group
Biological: Fluarix [NH 2006/07 season] — Single dose, intramuscular injection, Fluarix vaccine formulation recommended for the Northern Hemisphere 2006-2007 influenza season.
  Arms: Fluarix 2006/2007 Season Group
Biological: Fluarix [NH 2007/08 season] — Single dose, intramuscular injection, Fluarix vaccine formulation recommended for the Northern Hemisphere 2007-2008 influenza season.
  Arms: Fluarix 2007/2008 Season Group

SUMMARY:
This observer blind study is designed to compare the immune response of GSK Biologicals' influenza vaccine GSK576389A when administered using various presentations in adults aged 65 years and older. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
The study contains 6 parallel groups, stratified by two age groups: 65-74 years and ≥ 75 years and by two influenza vaccination histories: no influenza vaccination in the last 3 seasons and at least one influenza vaccination in the last 3 seasons.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female aged 65 years or older at the time of the vaccination.
* Written informed consent obtained from the subject.
* Free of an acute aggravation of the health status as established by clinical evaluation before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days prior to vaccination, or planned use during the study period.
* Administration of other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrolment in this study. Planned administration of a vaccine not foreseen by the study protocol up to Visit 2 after vaccination.
* Planned administration of an influenza vaccine other than the study vaccines during the entire study period.
* Vaccination against influenza since January 2007 (including the Northern Hemisphere NH 2006/2007 or NH 2007/08 influenza vaccine).
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the administration of the study vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* History of hypersensivity to a previous dose of influenza vaccine.
* History of allergy or reactions likely to be exacerbated by any component of the vaccine(s)
* Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by clinical evaluation or pre-existing laboratory screening tests.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first administration of the study vaccine or planned administration during the study.
* Any medical conditions in which intramuscular injections are contraindicated.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1596 (Actual)
Dates: Start 2007-09-20; Primary Completion 2007-11-01 (Actual); Study Completion 2007-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- GSK Investigational Site, Soeborg, Denmark
- GSK Investigational Site, Tartu, Estonia
- Norway (4):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Elverum
  - GSK Investigational Site, Hamar
  - GSK Investigational Site, Stavanger

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 110620 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110620 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110620 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110620 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110620 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110620 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110620 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two subjects enrolled in this study were not vaccinated and as such not accounted for under Started.
Period: Overall Study
Arm/Group | GSK576389A- 2006/2007 Season - 1 Container Group | GSK576389A - 2006/2007 Season - 2 Containers Group | Fluarix 2006/2007 Season Group | GSK576389A - 2007/2008 Season - 1 Container Group | GSK576389A - 2007/2008 Season - 2 Containers Group | Fluarix 2007/2008 Season Group
Started | 269 | 266 | 264 | 264 | 268 | 263
Completed | 267 | 265 | 263 | 264 | 267 | 261
Not Completed | 2 | 1 | 1 | 0 | 1 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK576389A- 2006/2007 Season - 1 Container Group | GSK576389A - 2006/2007 Season - 2 Containers Group | Fluarix 2006/2007 Season Group | GSK576389A - 2007/2008 Season - 1 Container Group | GSK576389A - 2007/2008 Season - 2 Containers Group | Fluarix 2007/2008 Season Group | Total
Number analyzed (Participants) | 269 | 266 | 264 | 264 | 268 | 263 | 1594
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.2 (5.56) | 73.0 (5.16) | 72.8 (5.06) | 73.3 (5.86) | 73.2 (5.72) | 73.0 (5.20) | 73.08 (5.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 149 | 150 | 145 | 152 | 153 | 900
  Male | 118 | 117 | 114 | 119 | 116 | 110 | 694

OUTCOME MEASURES:

1. Primary Outcome: Haemagglutination Inhibition (HI) Antibody Titers for the H1N1 Vaccine Strain
Description: Antibody titers were expressed as Geometric mean titers (GMTs). The H1N1 vaccine strains included A/New Caledonia and A/Solomon Islands antigens. A/New Caledonia vaccine strain was administered to both groups receiving the adjuvanted influenza vaccine GSK576389A for the Northern Hemisphere 2006/2007 influenza season. A/Solomon Islands vaccine strain was administered to both groups receiving the adjuvanted influenza vaccine GSK576389A for the Northern Hemisphere 2007/2008 influenza season.
Time Frame: At Days 0 and 21
Population: The analysis was performed on According-to-Protocol (ATP) immunogenicity cohort which included all evaluable subjects for whom data concerning immunogenicity were available. This primary outcome was assessed only on those groups receiving any of the GSK Bio's influenza vaccine GSK576389A formulations.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | GSK576389A- 2006/2007 Season - 1 Container Group | GSK576389A - 2006/2007 Season - 2 Containers Group | Fluarix 2006/2007 Season Group | GSK576389A - 2007/2008 Season - 1 Container Group | GSK576389A - 2007/2008 Season - 2 Containers Group | Fluarix 2007/2008 Season Group
Number analyzed (Participants) | 259 | 259 | 0 | 258 | 263 | 0
titer
  A/New Caledonia at Day 0 (N=259;259;0;0;0;0) | 37.9 [33.1 to 43.3] | 40.1 [34.7 to 46.4] |  | NA [NA to NA] — Subjects in this group were not analysed for A/New Caledonia vaccine strain as per protocol. | NA [NA to NA] — Subjects in this group were not analysed for A/New Caledonia vaccine strain as per protocol. |
  A/New Caledonia at Day 21 (N=259;259;0;0;0;0) | 130.8 [117.0 to 146.3] | 138.5 [123.2 to 155.8] |  | NA [NA to NA] — Subjects in this group were not analysed for A/New Caledonia vaccine strain as per protocol. | NA [NA to NA] — Subjects in this group were not analysed for A/New Caledonia vaccine strain as per protocol. |
  A/Solomon Islands at Day 0 (N=0;0;0;258;263;0) | NA [NA to NA] — Subjects in this group were not analysed for A/Solomon Islands vaccine strain as per protocol. | NA [NA to NA] — Subjects in this group were not analysed for A/Solomon Islands vaccine strain as per protocol. |  | 9.4 [8.4 to 10.5] | 9.0 [8.1 to 9.9] |
  A/Solomon Islands at Day 21 (N=0;0;0;258;263;0) | NA [NA to NA] — Subjects in this group were not analysed for A/Solomon Islands vaccine strain as per protocol. | NA [NA to NA] — Subjects in this group were not analysed for A/Solomon Islands vaccine strain as per protocol. |  | 82.0 [70.9 to 94.8] | 88.6 [76.4 to 102.7] |

2. Secondary Outcome: HI Antibody Titers Against Each of the Three Vaccine Strains for the Two Season Formulations
Description: Antibody titers were expressed as GMTs. The vaccine strains included A/New Caledonia or A/Solomon Islands, A/Wisconsin and B/Malaysia antigens. A/New Caledonia vaccine strain was administered to all groups receiving the Northern Hemisphere 2006/2007 influenza season vaccine formulations. A/Solomon Islands vaccine strain was administered to all groups receiving the Northern Hemisphere 2007/2008 influenza season vaccine formulations. A/Wisconsin and B/Malaysia vaccine strains were administered to all groups.
Time Frame: At Days 0 and 21
Population: The analysis was performed on According-to-Protocol (ATP) immunogenicity cohort which included all evaluable subjects for whom data concerning immunogenicity were available.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | GSK576389A- 2006/2007 Season - 1 Container Group | GSK576389A - 2006/2007 Season - 2 Containers Group | Fluarix 2006/2007 Season Group | GSK576389A - 2007/2008 Season - 1 Container Group | GSK576389A - 2007/2008 Season - 2 Containers Group | Fluarix 2007/2008 Season Group
Number analyzed (Participants) | 259 | 259 | 255 | 258 | 263 | 257
titer
  A/New Caledonia at Day 0 (N=259;259;255;0;0;0) | 37.9 [33.1 to 43.3] | 40.1 [34.7 to 46.4] | 35.3 [30.6 to 40.7] | NA [NA to NA] — Subjects in this group were not analysed for A/New Caledonia vaccine strain as per protocol. | NA [NA to NA] — Subjects in this group were not analysed for A/New Caledonia vaccine strain as per protocol. | NA [NA to NA] — Subjects in this group were not analysed for A/New Caledonia vaccine strain as per protocol.
  A/New Caledonia at Day 21 (N=259;259;255;0;0;0) | 130.8 [117.0 to 146.3] | 138.5 [123.2 to 155.8] | 114.7 [102.0 to 129.0] | NA [NA to NA] — Subjects in this group were not analysed for A/New Caledonia vaccine strain as per protocol. | NA [NA to NA] — Subjects in this group were not analysed for A/New Caledonia vaccine strain as per protocol. | NA [NA to NA] — Subjects in this group were not analysed for A/New Caledonia vaccine strain as per protocol.
  A/Solomon Islands at Day 0 (N=0;0;0;258;263;257) | NA [NA to NA] — Subjects in this group were not analysed for A/Solomon Islands vaccine strain as per protocol. | NA [NA to NA] — Subjects in this group were not analysed for A/Solomon Islands vaccine strain as per protocol. | NA [NA to NA] — Subjects in this group were not analysed for A/Solomon Islands vaccine strain as per protocol. | 9.4 [8.4 to 10.5] | 9.0 [8.1 to 9.9] | 8.5 [7.7 to 9.4]
  A/Solomon Islands at Day 21 (N=0;0;0;258;263;257) | NA [NA to NA] — Subjects in this group were not analysed for A/Solomon Islands vaccine strain as per protocol. | NA [NA to NA] — Subjects in this group were not analysed for A/Solomon Islands vaccine strain as per protocol. | NA [NA to NA] — Subjects in this group were not analysed for A/Solomon Islands vaccine strain as per protocol. | 82.0 [70.9 to 94.8] | 88.6 [76.4 to 102.7] | 61.0 [52.1 to 71.6]
  A/Wisconsin at Day 0 (N=259;259;255;258;263;257) | 47.7 [39.9 to 57.0] | 52.8 [44.1 to 63.2] | 53.3 [44.2 to 64.2] | 56.7 [47.7 to 67.5] | 52.8 [44.3 to 62.9] | 42.8 [35.8 to 51.2]
  A/Wisconsin at Day 21 (N=259;259;255;258;263;257) | 379.7 [328.5 to 439.0] | 409.9 [360.3 to 466.2] | 275.5 [241.6 to 314.3] | 399.9 [351.4 to 455.1] | 367.4 [322.9 to 418.2] | 178.9 [153.8 to 208.0]
  B/Malaysia at Day 0 (N=259;259;255;258;263;257) | 57.9 [50.4 to 66.6] | 59.5 [51.2 to 69.2] | 59.6 [50.9 to 69.7] | 68.0 [59.2 to 78.2] | 51.6 [44.8 to 59.6] | 54.3 [46.5 to 63.5]
  B/Malaysia at Day 21 (N=259;259;255;258;263;257) | 236.4 [212.6 to 262.9] | 213.8 [189.7 to 241.0] | 193.2 [170.0 to 219.5] | 253.6 [227.8 to 282.2] | 201.9 [180.0 to 226.6] | 180.5 [158.5 to 205.7]

3. Secondary Outcome: The Number of Subjects Seroconverted for HI Antibodies Against Each of the Three Vaccine Strains for the Two Season Formulations
Description: A seroconverted subject was defined as a subject who had either a pre-vaccination titer below 1:10 and a post-vaccination titer greater than or equal to 1:40 or a pre-vaccination titer greater than or equal to 1:10 and at least a 4-fold increase in post-vaccination titer. The vaccine strains included A/New Caledonia (for all groups receiving vaccine formulations for the Northern Hemisphere [NH] 2006/2007 influenza season) or A/Solomon Islands (for all groups receiving vaccine formulations for the NH 2007/2008 influenza season), A/Wisconsin and B/Malaysia antigens.
Time Frame: At Day 21
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | GSK576389A- 2006/2007 Season - 1 Container Group | GSK576389A - 2006/2007 Season - 2 Containers Group | Fluarix 2006/2007 Season Group | GSK576389A - 2007/2008 Season - 1 Container Group | GSK576389A - 2007/2008 Season - 2 Containers Group | Fluarix 2007/2008 Season Group
Number analyzed (Participants) | 259 | 259 | 255 | 258 | 263 | 257
Subjects
  A/New Caledonia strain (N=259;259;255;0;0;0) | 104 | 95 | 78 | NA — Subjects in this group were not analysed for A/New Caledonia vaccine strain as per protocol. | NA — Subjects in this group were not analysed for A/New Caledonia vaccine strain as per protocol. | NA — Subjects in this group were not analysed for A/New Caledonia vaccine strain as per protocol.
  A/Solomon Islands strain (N=0;0;0;258;263;257) | NA — Subjects in this group were not analysed for A/Solomon Islands vaccine strain as per protocol. | NA — Subjects in this group were not analysed for A/Solomon Islands vaccine strain as per protocol. | NA — Subjects in this group were not analysed for A/Solomon Islands vaccine strain as per protocol. | 177 | 192 | 161
  A/Wisconsin strain (N=259;259;255;258;263;257) | 177 | 188 | 128 | 171 | 173 | 109
  B/Malaysia strain (N=259;259;255;258;263;257) | 110 | 100 | 85 | 108 | 111 | 88

4. Secondary Outcome: HI Antibody Seroconversion Factors
Description: Seroconversion factors were defined as the fold increase in serum HI GMTs post-vaccination compared to Day 0. The vaccine strains included A/New Caledonia (for all groups receiving vaccine formulations for the Northern Hemisphere [NH] 2006/2007 influenza season) or A/Solomon Islands (for all groups receiving vaccine formulations for the NH 2007/2008 influenza season), A/Wisconsin and B/Malaysia antigens.
Time Frame: At Day 21
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | GSK576389A- 2006/2007 Season - 1 Container Group | GSK576389A - 2006/2007 Season - 2 Containers Group | Fluarix 2006/2007 Season Group | GSK576389A - 2007/2008 Season - 1 Container Group | GSK576389A - 2007/2008 Season - 2 Containers Group | Fluarix 2007/2008 Season Group
Number analyzed (Participants) | 259 | 259 | 255 | 258 | 263 | 257
fold increase
  A/New Caledonia strain (N=259;259;255;0;0;0) | 3.5 [3.0 to 4.0] | 3.5 [3.0 to 4.0] | 3.3 [2.8 to 3.8] | NA [NA to NA] — Subjects in this group were not analysed for A/New Caledonia vaccine strain as per protocol. | NA [NA to NA] — Subjects in this group were not analysed for A/New Caledonia vaccine strain as per protocol. | NA [NA to NA] — Subjects in this group were not analysed for A/New Caledonia vaccine strain as per protocol.
  A/Solomon Islands strain (N=0;0;0;258;263;257) | NA [NA to NA] — Subjects in this group were not analysed for A/Solomon Islands vaccine strain as per protocol. | NA [NA to NA] — Subjects in this group were not analysed for A/Solomon Islands vaccine strain as per protocol. | NA [NA to NA] — Subjects in this group were not analysed for A/Solomon Islands vaccine strain as per protocol. | 8.7 [7.5 to 10.2] | 9.9 [8.5 to 11.5] | 7.2 [6.1 to 8.4]
  A/Wisconsin strain (N=259;259;255;258;263;257) | 8.0 [6.7 to 9.4] | 7.8 [6.6 to 9.2] | 5.2 [4.3 to 6.3] | 7.0 [6.0 to 8.3] | 7.0 [5.9 to 8.3] | 4.2 [3.5 to 5.0]
  B/Malaysia strain (N=259;259;255;258;263;257) | 4.1 [3.5 to 4.7] | 3.6 [3.1 to 4.2] | 3.2 [2.8 to 3.8] | 3.7 [3.2 to 4.3] | 3.9 [3.4 to 4.5] | 3.3 [2.8 to 3.9]

5. Secondary Outcome: The Number of Subjects Seroprotected for HI Antibodies Against Each of the Three Vaccine Strains for the Two Season Formulations
Description: A seroprotected subject was defined as a subject with a serum HI titer greater than or equal to 1:40 that usually is accepted as indicating protection. The vaccine strains included A/New Caledonia (for all groups receiving vaccine formulations for the Northern Hemisphere [NH] 2006/2007 influenza season) or A/Solomon Islands (for all groups receiving vaccine formulations for the NH 2007/2008 influenza season), A/Wisconsin and B/Malaysia antigens.
Time Frame: At Days 0 and 21
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | GSK576389A- 2006/2007 Season - 1 Container Group | GSK576389A - 2006/2007 Season - 2 Containers Group | Fluarix 2006/2007 Season Group | GSK576389A - 2007/2008 Season - 1 Container Group | GSK576389A - 2007/2008 Season - 2 Containers Group | Fluarix 2007/2008 Season Group
Number analyzed (Participants) | 259 | 259 | 255 | 258 | 263 | 257
Subjects
  A/New Caledonia at Day 0 (N=259;259;255;0;0;0) | 160 | 163 | 156 | NA — Subjects in this group were not analysed for A/New Caledonia vaccine strain as per protocol. | NA — Subjects in this group were not analysed for A/New Caledonia vaccine strain as per protocol. | NA — Subjects in this group were not analysed for A/New Caledonia vaccine strain as per protocol.
  A/New Caledonia at Day 21 (N=259;259;255;0;0;0) | 252 | 246 | 239 | NA — Subjects in this group were not analysed for A/New Caledonia vaccine strain as per protocol. | NA — Subjects in this group were not analysed for A/New Caledonia vaccine strain as per protocol. | NA — Subjects in this group were not analysed for A/New Caledonia vaccine strain as per protocol.
  A/Solomon Islands at Day 0 (N=0;0;0;258;263;257) | NA — Subjects in this group were not analysed for A/Solomon Islands vaccine strain as per protocol. | NA — Subjects in this group were not analysed for A/Solomon Islands vaccine strain as per protocol. | NA — Subjects in this group were not analysed for A/Solomon Islands vaccine strain as per protocol. | 30 | 26 | 26
  A/Solomon Islands at Day 21 (N=0;0;0;258;263;257) | NA — Subjects in this group were not analysed for A/Solomon Islands vaccine strain as per protocol. | NA — Subjects in this group were not analysed for A/Solomon Islands vaccine strain as per protocol. | NA — Subjects in this group were not analysed for A/Solomon Islands vaccine strain as per protocol. | 202 | 215 | 187
  A/Wisconsin at Day 0 (N=259;259;255;258;263;257) | 169 | 174 | 172 | 180 | 171 | 158
  A/Wisconsin at Day 21 (N=259;259;255;258;263;257) | 252 | 257 | 249 | 255 | 259 | 239
  B/Malaysia at Day 0 (N=259;259;255;258;263;257) | 194 | 188 | 185 | 200 | 184 | 182
  B/Malaysia at Day 21 (N=259;259;255;258;263;257) | 255 | 253 | 249 | 257 | 260 | 246

6. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Adverse Events (AEs)
Description: Grade 3 ecchymosis, redness and swelling was greater than 100 millimeter (mm) i.e. >100mm and grade 3 pain was considerable pain at rest that prevented normal everyday activities. Any was occurrence of any local symptom regardless of their intensity grade. Any for ecchymosis, redness and swelling was >20mm.
Time Frame: During a 7-day follow-up period (Day 0-6) after vaccination
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented and symptom sheet completed.
Measure: Number; unit: Subjects
Arm/Group | GSK576389A- 2006/2007 Season - 1 Container Group | GSK576389A - 2006/2007 Season - 2 Containers Group | Fluarix 2006/2007 Season Group | GSK576389A - 2007/2008 Season - 1 Container Group | GSK576389A - 2007/2008 Season - 2 Containers Group | Fluarix 2007/2008 Season Group
Number analyzed (Participants) | 268 | 265 | 263 | 263 | 268 | 261
Subjects
  Any ecchymosis | 4 | 4 | 6 | 7 | 7 | 10
  Grade 3 ecchymosis | 1 | 0 | 0 | 1 | 0 | 1
  Any pain | 165 | 146 | 47 | 148 | 144 | 37
  Grade 3 pain | 0 | 2 | 0 | 1 | 3 | 0
  Any redness | 113 | 131 | 59 | 108 | 120 | 51
  Grade 3 redness | 19 | 27 | 4 | 19 | 24 | 0
  Any swelling | 52 | 53 | 13 | 53 | 49 | 18
  Grade 3 swelling | 4 | 6 | 0 | 0 | 5 | 0

7. Secondary Outcome: Duration of Solicited Local AEs
Description: Duration was defined as number of days with any grade of local symptoms.
Time Frame: During a 7-day follow-up period (Day 0-6) after vaccination
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented and symptom sheet completed only on subjects that reported the specific symptom.
Measure: Median (Full Range); unit: Days
Arm/Group | GSK576389A- 2006/2007 Season - 1 Container Group | GSK576389A - 2006/2007 Season - 2 Containers Group | Fluarix 2006/2007 Season Group | GSK576389A - 2007/2008 Season - 1 Container Group | GSK576389A - 2007/2008 Season - 2 Containers Group | Fluarix 2007/2008 Season Group
Number analyzed (Participants) | 165 | 146 | 58 | 148 | 144 | 50
Days
  Ecchymosis (N=4;4;5;7;7;10) | 3.0 [1.0 to 7.0] | 4.0 [3.0 to 5.0] | 6.0 [1.0 to 7.0] | 6.0 [3.0 to 7.0] | 3.0 [1.0 to 5.0] | 6.0 [1.0 to 7.0]
  Pain (N=165;146;47;148;144;37) | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0] | 3.0 [1.0 to 6.0] | 3.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0]
  Redness (N=113;131;58;108;120;50) | 3.0 [1.0 to 7.0] | 3.0 [1.0 to 7.0] | 3.0 [1.0 to 7.0] | 3.0 [1.0 to 7.0] | 4.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0]
  Swelling (N=52;53;12;53;49;18) | 3.0 [1.0 to 7.0] | 3.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0] | 2.0 [1.0 to 7.0] | 3.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0]

8. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General AEs
Description: Any temperature was defined as oral temperature greater than or equal to 38.0 degree centigrade i.e ≥38.0°C, grade 3 temperature was oral temperature ≥39.0°C. For other symptoms, any was defined as occurrence of any general symptom regardless of intensity grade or relation to vaccination and grade 3 was defined as a general symptom that prevented normal activity. Related was a general symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During a 7-day follow-up period (Day 0-6) after vaccination
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | GSK576389A- 2006/2007 Season - 1 Container Group | GSK576389A - 2006/2007 Season - 2 Containers Group | Fluarix 2006/2007 Season Group | GSK576389A - 2007/2008 Season - 1 Container Group | GSK576389A - 2007/2008 Season - 2 Containers Group | Fluarix 2007/2008 Season Group
Number analyzed (Participants) | 268 | 265 | 263 | 264 | 267 | 261
Subjects
  Any arthralgia | 58 | 36 | 19 | 39 | 30 | 20
  Grade 3 arthralgia | 3 | 0 | 1 | 1 | 1 | 1
  Related arthralgia | 57 | 36 | 16 | 39 | 30 | 19
  Any fatigue | 89 | 90 | 39 | 83 | 82 | 33
  Grade 3 fatigue | 4 | 3 | 0 | 4 | 1 | 0
  Related fatigue | 89 | 89 | 34 | 81 | 81 | 32
  Any headache | 76 | 67 | 26 | 62 | 58 | 27
  Grade 3 headache | 6 | 3 | 0 | 2 | 1 | 0
  Related headache | 73 | 64 | 23 | 62 | 58 | 23
  Any myalgia | 85 | 63 | 25 | 75 | 77 | 29
  Grade 3 myalgia | 1 | 0 | 1 | 0 | 2 | 0
  Related myalgia | 83 | 63 | 22 | 75 | 77 | 28
  Any nausea | 22 | 25 | 14 | 26 | 18 | 10
  Grade 3 nausea | 1 | 0 | 0 | 1 | 0 | 1
  Related nausea | 20 | 25 | 11 | 24 | 18 | 9
  Any shivering | 46 | 25 | 6 | 45 | 25 | 6
  Grade 3 shivering | 1 | 0 | 0 | 3 | 2 | 0
  Related shivering | 45 | 25 | 3 | 44 | 25 | 6
  Any temperature | 8 | 6 | 2 | 12 | 13 | 2
  Grade 3 temperature | 1 | 1 | 0 | 1 | 1 | 0
  Related temperature | 8 | 6 | 1 | 12 | 13 | 1

9. Secondary Outcome: Duration of Solicited General AEs
Description: Duration was defined as number of days with any grade of general symptoms.
Time Frame: During a 7-day follow-up period (Day 0-6) after vaccination
Population: as for outcome 7
Measure: Median (Full Range); unit: Days
Arm/Group | GSK576389A- 2006/2007 Season - 1 Container Group | GSK576389A - 2006/2007 Season - 2 Containers Group | Fluarix 2006/2007 Season Group | GSK576389A - 2007/2008 Season - 1 Container Group | GSK576389A - 2007/2008 Season - 2 Containers Group | Fluarix 2007/2008 Season Group
Number analyzed (Participants) | 89 | 90 | 39 | 83 | 82 | 33
Days
  Arthralgia (N=58;36;19;39;30;20) | 2.0 [1.0 to 7.0] | 1.5 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0] | 3.0 [1.0 to 7.0]
  Fatigue (N=89;90;39;83;82;33) | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 1.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Headache (N=76;67;26;62;58;27) | 1.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 1.5 [1.0 to 7.0] | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 6.0] | 2.0 [1.0 to 7.0]
  Myalgia (N=85;63;25;75;77;29) | 2.0 [1.0 to 6.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Nausea (N=22;25;14;26;18;10) | 1.0 [1.0 to 5.0] | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 3.0] | 1.5 [1.0 to 4.0]
  Shivering (N=46;25;6;45;25;6) | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 5.0] | 1.0 [1.0 to 5.0] | 1.0 [1.0 to 2.0]
  Temperature (N=4;4;1;7;9;0) | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 3.0 [3.0 to 3.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 4.0] | NA [NA to NA] — Information on duration of fever was missing from these subject's symptom sheets

10. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited AEs
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination. Grade 3 was an event that prevented normal activities and related was defined as an unsolicited AE assessed by the investigator to be causally related to the study vaccination.
Time Frame: During a 21-day follow-up period (Day 0-20) after vaccination
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | GSK576389A- 2006/2007 Season - 1 Container Group | GSK576389A - 2006/2007 Season - 2 Containers Group | Fluarix 2006/2007 Season Group | GSK576389A - 2007/2008 Season - 1 Container Group | GSK576389A - 2007/2008 Season - 2 Containers Group | Fluarix 2007/2008 Season Group
Number analyzed (Participants) | 269 | 266 | 264 | 264 | 268 | 263
Subjects
  Any AE(s) | 43 | 39 | 36 | 45 | 53 | 29
  Grade 3 AE(s) | 2 | 1 | 0 | 3 | 2 | 1
  Related AE(s) | 22 | 21 | 11 | 28 | 30 | 12

11. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Medically Significant Conditions (MSCs)
Description: MSCs were defined as an AEs with a medically-attended visit (MAE) i.e. prompting emergency room (ER) visits, hospitalizations or physician visits and that were not routine visits for physical examination or vaccination. Any MSC was defined as at least one MSC experienced. Grade 3 was a MSC that prevented normal activities and related was defined as a MSC assessed by the investigator to be causally related to the study vaccination.
Time Frame: During a 21-day follow-up period (Day 0-20) after vaccination
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | GSK576389A- 2006/2007 Season - 1 Container Group | GSK576389A - 2006/2007 Season - 2 Containers Group | Fluarix 2006/2007 Season Group | GSK576389A - 2007/2008 Season - 1 Container Group | GSK576389A - 2007/2008 Season - 2 Containers Group | Fluarix 2007/2008 Season Group
Number analyzed (Participants) | 269 | 266 | 264 | 264 | 268 | 263
Subjects
  Any MSC(s) | 7 | 4 | 11 | 5 | 11 | 9
  Grade 3 MSC(s) | 0 | 1 | 0 | 1 | 1 | 1
  Related MSC(s) | 1 | 0 | 1 | 0 | 4 | 2

12. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: During a 21-day follow-up period (Day 0-20) after vaccination
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | GSK576389A- 2006/2007 Season - 1 Container Group | GSK576389A - 2006/2007 Season - 2 Containers Group | Fluarix 2006/2007 Season Group | GSK576389A - 2007/2008 Season - 1 Container Group | GSK576389A - 2007/2008 Season - 2 Containers Group | Fluarix 2007/2008 Season Group
Number analyzed (Participants) | 269 | 266 | 264 | 264 | 268 | 263
Subjects
  Any SAE(S) | 2 | 0 | 0 | 2 | 0 | 1
  Related SAE(s) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events were assessed from day 0 to day 20. Systematically assessed frequent adverse events (AEs) and non-systematically assesed frequent AEs were assessed during 7 day and 21 day post vaccination period respectively.
Description: For the systematically assessed other (non-serious) adverse events, the number of participants at risk included those from Total Vaccinated cohort who had the symptom sheet completed.
Arm/Group | GSK576389A- 2006/2007 Season - 1 Container Group | GSK576389A - 2006/2007 Season - 2 Containers Group | Fluarix 2006/2007 Season Group | GSK576389A - 2007/2008 Season - 1 Container Group | GSK576389A - 2007/2008 Season - 2 Containers Group | Fluarix 2007/2008 Season Group
Serious Adverse Events (participants affected / at risk) | 2/269 | 0/266 | 0/264 | 2/264 | 0/268 | 1/263
Other Adverse Events (participants affected / at risk) | 233/269 | 224/266 | 145/264 | 224/264 | 219/268 | 138/263
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK576389A- 2006/2007 Season - 1 Container Group (N=269) | GSK576389A - 2006/2007 Season - 2 Containers Group (N=266) | Fluarix 2006/2007 Season Group (N=264) | GSK576389A - 2007/2008 Season - 1 Container Group (N=264) | GSK576389A - 2007/2008 Season - 2 Containers Group (N=268) | Fluarix 2007/2008 Season Group (N=263)
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | GSK576389A- 2006/2007 Season - 1 Container Group (N=269) | GSK576389A - 2006/2007 Season - 2 Containers Group (N=266) | Fluarix 2006/2007 Season Group (N=264) | GSK576389A - 2007/2008 Season - 1 Container Group (N=264) | GSK576389A - 2007/2008 Season - 2 Containers Group (N=268) | Fluarix 2007/2008 Season Group (N=263)
Pain (General disorders) | 165/268 | 146/265 | 47/263 | 148/263 | 144 | 37/261
Redness (General disorders) | 113/268 | 131/265 | 59/263 | 108/263 | 120 | 51/261
Swelling (General disorders) | 52/268 | 53/265 | 13/263 | 53/263 | 49 | 18/261
Arthralgia (General disorders) | 58/268 | 36/265 | 19/263 | 39 | 30/267 | 20/261
Fatigue (General disorders) | 89/268 | 90/265 | 39/263 | 83 | 82/267 | 33/261
Headache (General disorders) | 76/268 | 67/265 | 26/263 | 62 | 58/267 | 27/261
Myalgia (General disorders) | 85/268 | 63/265 | 25/263 | 75 | 77/267 | 29/261
Nausea (General disorders) | 22/268 | 25/265 | 14/263 | 26 | 18/267 | 10/261
Shivering (General disorders) | 46/268 | 25/265 | 6/263 | 45 | 25/267 | 6/261
Injection site pruritus (General disorders) | 12 | 14 | 7 | 13 | 15 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.